CLINICAL TRIAL: NCT00230880
Title: Randomized Trial of an Intervention to Impact Contraceptive Behavior, Unintended Pregnancy, and STIs Among Adolescent Females Receiving Family Planning Clinic Services
Brief Title: The Young Woman's Reach Project: Trial of an Intervention to Impact Contraceptive Behavior, Unintended Pregnancy, and Sexually Transmitted Infections (STIs) Among Adolescent Females
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: ETR Associates (Other); William and Flora Hewlett Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: OSR# 04038166
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Contraceptive Behavior; Sexually Transmitted Diseases
Keywords: Contraception behavior; Condoms; Unsafe sex; Pregnancy unwanted; Adolescent pregnancy; Condom use; Unprotected sex; Unintended pregnancy
MeSH Terms: conditions — Contraception Behavior; Sexually Transmitted Diseases; Unsafe Sex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): follow-up phone counseling
  Interventions: Behavioral: follow-up phone counseling
- Control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: follow-up phone counseling — 9 calls over 12 months
  Other Names: Intense phone follow-up using motivational interviewing
  Arms: Treatment

SUMMARY:
The New Generation Health Center/University of California, San Francisco (UCSF) will implement an intervention to impact contraceptive behavior and reduce unintended pregnancy and sexually transmitted infections (STIs) among adolescent females who receive services at the New Generation Health Center (NGHC)/UCSF in San Francisco. Study subjects will be randomized into either standard reproductive health services or standard services plus follow-up motivational counseling telephone calls. Outcomes will be evaluated by ETR (Education, Training, Research)Associates, who will conduct follow-up surveys with all study participants at baseline, 6 months, 12 months and 18 months.

DETAILED DESCRIPTION:
The United States has one of the highest teen pregnancy rates of any western industrialized nation. In 1999, the last year for which state pregnancy data are available, California had the seventh highest pregnancy rate in the country. Within San Francisco, the Mission and Bayview Hunters Point districts have rates that are almost three times and two times higher than the state average respectively. In addition to high rates of unintended pregnancy, residents in the Bayview Hunters Point district experience STI transmission rate much higher than that of other neighborhoods.

Currently there is very little research on the impact of different types of reproductive health clinic protocols on adolescent contraceptive use. Different outcomes have been found in the few studies that do exist on this topic. Hercog-Baron found that follow-up phone calls did not affect contraceptive use; however, explained that most youth stopped using contraception after the first three months of supply had run out and no calls were made beyond that time-frame. Authors suggested that the intervention may be more effective with a longer duration of follow-up. Alternatively, another study reported that their program substantially reduced teen pregnancy rates over time. Although the intervention had many components, the authors reported that the staff credited the positive relationships they created between the health educator and each student, and the frequent reminders contributed to the reduction in sexual risk-taking and pregnancy.

A review by Miller and Sanchez concluded that the following seven elements of brief interventions induced positive change in a variety of health areas:

1. feedback and counseling on personal risk,
2. emphasis on personal responsibility for change,
3. clear message about behavior change,
4. a menu of behavior change options,
5. therapist/counselor empathy,
6. facilitation of client self-efficacy and
7. use of a "motivational interviewing style".

To the extent feasible, these elements will be incorporated into the Project REACH phone calls. Although there is very little data available in this area, the studies summarized above suggest that multiple contacts over time, even though brief, can have an impact.

The NGHC will improve its reproductive health services by expanding current services to include a series of follow-up phone calls. The main purpose of these calls will be to assess how well patients are doing, to discuss any questions or problems they have had with their methods, and to enforce the four main messages:

1. encourage condom use,
2. encourage patients to return to the clinic for hormonal methods of contraception if they are likely to remain sexually active or want to change their method of contraception,
3. get STI tested annually or if at risk and
4. use the clinic as a resource and return for reproductive health needs.

Clinics in San Francisco and around the country do not know whether conducting follow-up calls improves contraception compliance, increases STI testing or decreases unintended pregnancy. This study will significantly increase the field's knowledge of the feasibility and impact of conducting follow-up calls with youth over an extended period of time after they come to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Attending a family planning clinic visit
* At risk for unintended pregnancy (using no contraceptive method, using condoms for contraception, or not using a hormonal contraceptive method continuously for the last 3 months)

Exclusion Criteria:

* Pregnant
* Using a hormonal contraceptive method continuously for the last 3 months
* Not willing to be contacted by phone for the intervention.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 800 (Actual)
Dates: Start 2005-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Contraceptive use at time of last sexual intercourse | 18 months

SECONDARY OUTCOMES:
Unintended pregnancy | 18 months
Sexually transmitted infections | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Tina R Raine-Bennett, MD, MPH, Principal Investigator — University of California, San Francisco; Doug Kirby, PhD, Principal Investigator — ETR Associates
Locations (1):
- New Generation Health Center/UCSF, San Francisco, California, United States